CLINICAL TRIAL: NCT01863134
Title: Clinical Effects of Eptifibatide Administration in High Risk Patients Presenting With Non-ST Segment Elevation Acute Coronary Syndrome (NSTE-ACS) Requiring Urgent Coronary Artery Bypass Graft Surgery in Short- and Long-Term Follow-up
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Miroslaw Wilczynski, MD, PhD, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2 P05C 023 27
Record Dates: First submitted 2013-05-18; First posted 2013-05-27 (Estimated); Results first posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-08

CONDITIONS: Non ST Elevation Myocardial Infarction
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Eptifibatide; Weights and Measures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eptifibatide (Experimental): Patients were given a bolus of eptifibatide (Integrillin; 180µg/kg of body weight) and an intravenous infusion of 2 µg/kg/min followed by acetylsalicylic acid (150mg orally daily until the day of the procedure) and enoxaparin (1mg/kg subcutaneous - with the last dose 12 hours before surgery).
  Interventions: Drug: Eptifibatide
- Placebo (Placebo Comparator): Patients were given placebo infusion (0,9% Natrium Chloride) and an intravenous infusion of 2 µg/kg/min followed by acetylsalicylic acid (150mg orally daily until the day of the procedure) and enoxaparin (1mg/kg subcutaneous - with the last dose 12 hours before surgery).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eptifibatide
  Other Names: In the active treatment arm patients were additionally treated with eptifibatide (Integrillin; 180µg/kg of body weight) at an infusion rate 2 µg/kg/min
  Arms: Eptifibatide
Drug: Placebo
  Arms: Placebo

SUMMARY:
1. INTRODUCTION

   Through last couple of years the number of patients treated for acute coronary event without persistent ST segment elevation in ECG has been growing.

   This is probably an effect of improving diagnostics of myocardial infraction without persistent ST segment elevation in ECG, due to routine Troponin serum level evaluation and better primary prevention.

   This fact makes the search for the optimal treatment for patients with acute coronary event without persistent ST segment elevation in ECG, including both patients intended for pharmacological and invasive treatment percutaneous coronary intervention (PCI) or coronary artery byppass grafting (CABG).

   Patients undergoing invasive treatment for acute coronary event, have higher risk rate, than those with stabile angina pectoris.

   The authors of this study want to evaluate, whether the proportional use of platelet GP IIb/IIIa receptor antagonist - eptifibatide in patients undergoing CABG results in improvement of short-, and long time results in those patients.

   Eptifibatide ( Integrilin) a cyclic heptapeptide antagonist of the GP IIb/IIIa integrin receptor, is an intravenous antagonist with rapid onset and short half-life.
2. STUDY RATIONALE

The notion acute coronary syndrome (ACS) includes several clinical situations, such a unstable coronary artery disease, non-Q wave myocardial infarction and Q wave myocardial infarction.

On the basis of 12-lead ECG, patients with acute coronary syndrome (ACS) can be divided into two groups: with and without ST segment elevation.

Another stratification factor in patients with ACS, especially these without ST elevation is evaluation of biochemical markers of myocardial necrosis, such as Troponins (TnI, TnT) and creatinine kinase isoenzymes (CK-MB). Serum concentrations of these markers allow to distinguish myocardial infarction (elevation of markers' concentration) from unstable coronary artery disease.

All ACS have common etiopathogenesis which is plaque rupture, thrombus formation in the lumen of coronary artery.

Platelets are the key factor in this process. Platelets by means of their collagen and von Willebrand factor glycoprotein receptors bind to damaged artery wall. Simultaneously many factors cause platelet activation, which leads to changes in their shape, release of intraplatelet components and activation of fibrinogen-binding glycoprotein receptors IIb/IIIa (GP IIb/IIIa). Activated form of GP IIb/IIIa binds to GP IIb/IIIa of another platelet by means of fibrinogen molecule. Fibrinogen molecules form stable bridges between platelets. This process is referred to as aggregation, and leads to clot formation, which is further stabilized by fibrine fibres.

In this way the intravascular thrombus is formed, which after totally occluding the arterial lumen causes acute ischemia of the relevant region of myocardium and subsequently its infarction.

The key role of GP IIa/IIIb in the process of platelet clot formation has important therapeutic consequences. By now several specific (direct) and non-specific (indirect) antagonists of GP IIb/IIIa have been developed.

There are indirect antagonists as acetylsalicylic acid, ticlopidine and clopidogrel and direct antagonists as abciximab, tirofiban and eptifibatide Additionally also anticoagulants (heparin, LMWH - low molecular weight heparin) have antiplatelet properties by inhibiting thrombin production.

Clinical studies performed all over the world have proven the efficacy and safety of three agents from the GP Iia/IIIb group: abciximab, tirofiban and eptifibatide.

In several big clinical studies (EPIC, EPILOG, EPISTENT, ESPRIT, CAPTURE, PURSUIT, PRISM-PLUS, TACTICS-TIMI 18) the high efficacy of these drugs was showed in patients with ACS without ST segment elevation undergoing mainly percutaneous transluminal coronary angiography (PTCA) and stenting. The use of GP IIa/IIIb antagonists in this group of patients significantly reduces the death and myocardial infarction (MI) rate during early as well as late follow-up period. Moreover, last observations indicate, that the biggest benefit from such therapeutic strategy is observed in high risk patients; those with diabetes, high troponin levels and ECG changes.

During last years, there is an increase in frequency of ACS without ST segment elevation. This is probably due to improved diagnostics of MI without ST elevation basing on routine troponin evaluation, but also thanks to better primary prevention.

Therefore determining an optimal therapeutic strategy for patients with ACS without ST segment elevation remains a crucial issue.

It concerns patients qualified to medical treatment as well as those qualified to invasive procedures (PTCA or CABG).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a typical anginal pain lasting at least 20 min., but no longer than 24h.
* ECG confirming ischaemia
* ST segment depression >= 1,0 mm in at least 2 leads, or,
* negative T waves >= 2,0 mm in at least 2 leads.
* Positive troponin I (TnI).
* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent and/or parent or legal guardian must have signed a written informed consent.
* Subjects must be ≥ 21 year of age, of either sex and any race.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed IUD - intrauterine device, condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Subjects must be free of any clinically significant disease that would interfere with study evaluations (see exclusion criteria).
* Subjects must understand and be able to adhere to the dosing and visit schedules, and agree to record concomitant medications and adverse events.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications.
* Subjects who have used any investigational product within 30 days prior to enrollment.
* Subjects who have the following clinical conditions are excluded:

Patients with:

* Angina lasting longer than 24h.
* ST segment elevation - Pardy wave
* age over 75 years
* history of revascularization procedure during last 6 months (PTCA, CABG)
* chronic heart failure (NYHA III or IV) during pre-hospitalization period
* history of bleeding from gastrointestinal tract or genitourinary system during last 30 days
* history of intracranial lesions or stroke
* history of major surgery or trauma during last 6 weeks
* history of hemorrhagic diathesis
* thrombocytopenia < 100 000/mm3
* anticoagulant therapy with INR>2,0
* significant hepatic failure
* significant renal failure with serum creatinine>2,0 mg%
* elevated blood pressure: SBP>200mmHg and/or DBP>110mmHg despite the antihypertensive treatment
* allergy to drugs or any therapeutic agent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miroslaw Wilczynski, MD, PhD, Principal Investigator — Medical University of Silesia
Locations (6):
- Albert Einstein College of Medicine, New York, New York, United States
- Poland (5):
  - First Department of Cardiac Surgery, Medical University of Silesia, Katowice, Silesian Voivodeship
  - Center for Cardiovascular Research and Development, American Heart of Poland, Katowice
  - Department of Internal Medicine and Clinical Pharmacology, Katowice
  - First Department of Cardiology, Medical University of Silesia, Katowice
  - Division of Molecular Biology and Clinical Genetics, Jagiellonian University Medical College, Krakow

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four clinical centers located within a radius of 50km of the reference center were selected for the study. From 2005 to 2010 a total of 140 patients presenting with NSTE-ACS not eligible for PCI were enrolled to the study. All CABG procedures were performed at 1st Department of Cardiac Surgery, Silesian Medical University in Katowice.
Groups:
- Eptifibatide: Patients were given a bolus of eptifibatide (Integrillin; 180µg/kg of body weight) and an intravenous infusion of 2 µg/kg/min followed by acetylsalicylic acid (150mg PO daily until the day of the procedure) and enoxaparin (1mg/kg SC - with the last dose 12 hours before surgery).
- Placebo: Patients were given placebo infusion (0,9% Natrium Chloride) and an intravenous infusion of 2 µg/kg/min followed by acetylsalicylic acid (150mg PO daily until the day of the procedure) and enoxaparin (1mg/kg SC - with the last dose 12 hours before surgery).
Period: Overall Study
Arm/Group | Eptifibatide | Placebo
Started | 72 | 68
Completed | 72 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Control Group: In the control group patients were given identical doses of acetylsalicylic acid and enoxaparin followed by a placebo infusion of saline in lieu of the GPIIb/IIIa inhibitor.
- Eptifibatide: In the treatment group patients were given a bolus of eptifibatide (Integrillin; 180µg/kg of body weight) and an intravenous infusion of 2 µg/kg/min followed by acetylsalicylic acid (150mg PO daily until the day of the procedure) and enoxaparin (1mg/kg SC - with the last dose 12 hours before surgery). The minimal and maximal periods of eptifibatide infusion were established at 12 and 48 hours respectively.
- Total: Total of all reporting groups
Arm/Group | Placebo/Control Group | Eptifibatide | Total
Number analyzed (Participants) | 68 | 72 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 61 | 119
  >=65 years | 10 | 11 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 63.60 (8.32) | 62.47 (10.41) | 63.01 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 49 | 51 | 100
Region of Enrollment [Number; unit: participants]
  Poland | 68 | 72 | 140

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac and Cerebrovascular Events (MACCE)
Description: MACCE was defined as combined death, nonfatal myocardial infarction, cerebrovascular event (stroke) and the need for re-hospitalization due to recurrent ischemia up to 12 months follow-up
Time Frame: Up to 12 month
Measure: Number; unit: Percentage of study group
Arm/Group | Placebo | Eptifibatide
Number analyzed (Participants) | 68 | 72
Percentage of study group | 35.3 | 13.8

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Death up to 12 Months
Arm/Group | Eptifibatide | Placebo
Serious Adverse Events (participants affected / at risk) | 2/72 | 7/68
Other Adverse Events (participants affected / at risk) | 3/72 | 9/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptifibatide (N=72) | Placebo (N=68)
Death up to 12 Months (General disorders) | 2 (2) | 7 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptifibatide (N=72) | Placebo (N=68)
Pulmonary infection (Infections and infestations) | 3 (3) | 5 (5)
Delirium (Nervous system disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes